CLINICAL TRIAL: NCT03360318
Title: Brace Versus Casting in Pediatric Radial Head Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, pengzhang, Department of orthopaedics and trauma, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CSG-03qtd
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Radial Fracture
Keywords: pediatric; elbow fractures; management
MeSH Terms: conditions — Radius Fractures; Elbow Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elbow cast (Active Comparator): Device: Elbow cast
  Interventions: Device: elbow cast
- Removable elbow brace (Experimental): Device: Removable elbow brace
  Interventions: Device: Removable elbow brace

INTERVENTIONS:
Device: elbow cast — elbow cast
  Arms: Elbow cast
Device: Removable elbow brace — Removable elbow brace
  Arms: Removable elbow brace

SUMMARY:
Commare the pain and function of Brace Versus Casting in Pediatric Radial Head Fractures after 1 month

DETAILED DESCRIPTION:
Radial Head Fractures are common injury in children. In this study, healthy children with Mason type I or II radial head fractures are planned to be included.

Outcome Measures: The primary outcome measure will be an assessment of functional daily activities as measured by the MAYO score at four weeks post injury. Secondary outcomes will include an assessment of pain scores using VAS.

Sample Size and Analysis: Assuming a standard deviation of 10%, alpha = 0.05, beta = 0.2 and 10% dropout rate yields a sample size of 150 patients. Secondary analyses will include Fisher's Exact test to compare proportions of children with full range of motion of the injured ankle at four weeks and with full baseline activity level at four months, and the area under the curve of a pain-time profile curve will be compared using a Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

5 to 18 years of age with one of the following fracture Undisplaced Maoson types I and II fractures of the radial head

Exclusion Criteria:

The diagnosis of elbow sprain or contusion; they occur primarily in adolescents with closed epiphyseal plates.

All open fractures which require surgical debridement. All children at risk for pathological fractures such as those with congenital or acquired generalized bony disease.

Congenital anomalies of the elbow. Patients with coagulopathies. Multisystem trauma and multiple fractures of the same or opposite limb. Patients cognitively and developmentally delayed with inability to express pain and/or difficult assessment of baseline activity level.

Injuries greater than 72 hours old. Past history of surgery or closed reduction of the same elbow within the last 6 months or ankle trauma of the same ankle within 3 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02-02 (Estimated); Primary Completion 2019-02-05 (Estimated); Study Completion 2019-02-05 (Estimated)

PRIMARY OUTCOMES:
Mayo score | 1 month
  Functional outcome as measured by the Mayo score at 4 weeks from the time of the initial injury

SECONDARY OUTCOMES:
pain | 1 month
  VAS score

CONTACTS AND LOCATIONS:
Overall Officials: peng zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China